CLINICAL TRIAL: NCT04393753
Title: A Phase II, Open Label Study to Investigate the Efficacy and Safety of Domatinostat in Combination With Avelumab in Patients With Advanced Unresectable/Metastatic Merkel Cell Carcinoma Progressing on Anti-PD-(L)1 Antibody Therapy
Brief Title: Domatinostat in Combination With Avelumab in Patients With Advanced Merkel Cell Carcinoma Progressing on Anti-PD-(L)1
Acronym: MERKLIN2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 4SC AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4SC-202-3-2018; 2018-004788-30 (EudraCT Number)
Record Dates: First submitted 2020-05-12; First posted 2020-05-19 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — domatinostat; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- domatinostat and avelumab (Experimental): Single arm study of Domatinostat tablets in combination with avelumab infusion
  Interventions: Drug: domatinostat in combination with avelumab

INTERVENTIONS:
Drug: domatinostat in combination with avelumab — domatinostat tablets and avelumab infusion

SUMMARY:
This phase II trial studies how well domatinostat (4SC-202) works in combination with avelumab in adult patients with advanced unresectable and/or metastatic Merkel Cell Carcinoma that have progressed on a previous therapy with an anti-PD-(L)1 antibody

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Merkel Cell Carcinoma (MCC)
* ECOG performance status ≤ 1
* MCC in an advanced, unresectable stage III or metastatic stage IV (includes patients who refused surgical resection or are not eligible for such surgical resection)
* Progressing on previous anti-PD-(L)1 antibody monotherapy within the last 12 weeks before planned first administration of study medication

Exclusion Criteria:

* History of serious anti-PD-(L)1 therapy-related adverse reactions prohibiting further avelumab treatment
* More than one line of previous systemic anti-neoplastic therapy other than anti-PD-(L)1 antibody monotherapy
* Palliative radiation therapy of single lesions within 2 weeks before planned administration of study medication
* Presence of significant active or chronic disease (infections, immunodeficiencies, cardiovascular, psychiatric disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months
  Objective Response Rate (ORR) defined as the percentage of patients having a confirmed CR or PR according to RECIST v1.1

SECONDARY OUTCOMES:
Durable Response Rate (DRR) | up to 24 months
  Durable Response Rate (DRR), defined as the percentage of patients having a RECIST v1.1 response lasting ≥ 6 months
Duration of Response (DoR) | up to 24 months
  Duration of Response (DoR), defined as the time from an initial objective response (CR or PR) according to RECIST v1.1 until disease progression or death due to any cause
Disease Control Rate (DCR) | up to 24 months
  Disease Control Rate (DCR), defined as the proportion of patients with either an objective response (CR, PR) or stable disease (SD) according to RECIST v1.1.
Durable Disease Control Rate (dDCR) | up to 24 months
  Durable Disease Control Rate (dDCR), defined as the percentage of patients having a RECIST v1.1 disease control lasting ≥ 6 months
Best Overall response (BOR) | up to 24 months
  Best Overall response (BOR), defined as the best response (PD, SD, PR, CR) according to RECIST v1.1 over the course of a patient's participation in the study, assessed up to 2 years
Progression Free Survival (PFS) | up to 24 months
  Progression Free Survival (PFS), defined as the time from first dosing (Day +1) to the date of PD or death from any cause (whichever comes first)
PFS Rate | up to 24 months
  PFS Rate, defined as the percentage of patients without PD at 6 and 12 months after first administration of study drug
Overall Survival (OS) | up to 36 months
  Overall Survival (OS), defined as the time from the first administration of study medication until death due to any cause
OS Rate | up to 12 months
  OS Rate, defined as the percentage of patients alive at 6 and at 12 months after first administration of study drug
Safety and Tolerability | up to 24 months
  Safety and Tolerability of the study medication (determined by number, frequency, duration and severity of AEs using CTCAE v5.0, physical examination, laboratory tests, vital signs, and ECGs)
Health related Quality of Life (HrQoL) | up to 24 months
  The impact of treatment on the patient's QoLwill be assessed with the questionnaires "Functional Assessment of Cancer Therapy - Melanoma (FACT-M)" where QoL is assessed on a scale 0-240 (higher score means better status of health), with "EQ-5D-5L" which is a multi attribute utility instrument for measuring health-related QoL as EQ5D index with a score 0-1 (higher score means better status of health) and with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) with a score 0-100 per subscale (n=9 per item (n=6), higher score means better QoL.
Plasma concentration of domatinostat and avelumab | up to 48 weeks
  Single trough values of domatinostat and avelumab at pre-defined time points
Avelumab anti-drug antibodies (ADA) | up to 48 weeks
  Avelumab anti-drug antibodies (ADA)

CONTACTS AND LOCATIONS:
Locations (22):
- UZ Leuven, Leuven, Belgium
- France (4):
  - Bordeaux Hôpital Saint Andre, Bordeaux
  - Hôpital Ambroise Paré - Boulogne-Billancourt, Boulogne-Billancourt
  - CHU Nantes - Hotel Dieu, Nantes
  - Hôpital Saint-Louis, Paris
- Germany (10):
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Dresden, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Technische Universität München, München
  - Universitätsklinikum Tübingen, Tübingen
- Italy (4):
  - Instituto Tumori Giovanni Paolo II IRCCS Ospedale Oncologico Bari, Bari
  - Istituto Nazionale Tumori Fondazione G.Pascale, Naples
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Fondazione del Piemonte per l'Oncologia, Torino
- Netherlands (2):
  - Netherlands Cancer Institute Amsterdam, Amsterdam
  - Academic Hospital Maastricht, Maastricht
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No